CLINICAL TRIAL: NCT06726200
Title: A Randomized Controlled Trial Examining Extended-Release Injectable Buprenorphine in Those Who Use High Potency Synthetic Opioids
Brief Title: A Clinical Trial Comparing Buprenorphine Formulations for High Potency Synthetic Opioid Use
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rachel R. Luba (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Rachel R. Luba, Associate Research Scientist, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAV2503; K23DA057392-01A1 (NIH)
Record Dates: First submitted 2024-12-03; First posted 2024-12-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Naloxone; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Injectable Buprenorphine (Experimental): Long-Acting Injectable Buprenorphine administered after participants receive and tolerate a single 4/1 mg sublingual buprenorphine/naloxone dose
  Interventions: Drug: Buprenorphine Injection
- Sublingual Buprenorphine/Naloxone (Active Comparator): Titration onto sublingual buprenorphine/naloxone (standard of care)
  Interventions: Drug: Buprenorphine + naloxone (Suboxone)

INTERVENTIONS:
Drug: Buprenorphine + naloxone (Suboxone) — Participants randomized to sublingual buprenorphine naloxone will initiate treatment based on clinical guidelines/standard of care
  Arms: Sublingual Buprenorphine/Naloxone
Drug: Buprenorphine Injection — Participants randomized to injectable buprenorphine naloxone will receive a 300mg injection after receiving/tolerating a single 4/1 mg sublingual buprenorphine/naloxone dose
  Arms: Injectable Buprenorphine

SUMMARY:
The goal of this clinical trial is to compare buprenorphine formulations (sublingual buprenorphine versus long-acting injectable buprenorphine) for treating opioid use disorder among individuals who use fentanyl and/or other high potency synthetic opioids. Individuals aged 18-65 will be eligible for enrollment. The main questions it aims to answer are:

Are there differences in frequency of drug use after individuals start treatment with sublingual buprenorphine compared to injectable buprenorphine?

Are there differences in rates of sustained relapse after individuals start treatment with sublingual buprenorphine compared to injectable buprenorphine?

Investigators also seek to understand and explore:

How factors like body fat, body weight, and quantity of fentanyl use before treatment influence treatment outcomes.

How blood levels of buprenorphine and its metabolite norbuprenorphine early on in treatment may influence treatment outcomes.

How factors like craving and opioid withdrawal symptoms influence treatment outcomes.

Participants will:

Complete a brief overnight hospital stay in an inpatient research unit. This hospital stay will enable participants to start treatment with either sublingual buprenorphine or injectable buprenorphine.

Provide blood and urine samples while on the inpatient unit and at follow up.

Complete in-person follow up visits at 1-, 2-, 3- and 4-weeks after leaving the hospital to measure drug use, craving, withdrawal, quality of life, and physical health.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65
* Voluntarily seeking treatment for opioid use disorder (OUD)
* Consistent use of fentanyl or other high potency synthetic opioids
* Meets DSM-5 criteria for OUD with at least moderate severity
* Able to provide written informed consent in English and willing to comply with study procedures

Exclusion Criteria:

* Meets DSM-5 criteria for another substance use disorder as the primary diagnosis
* Has an active, unmanaged psychiatric condition that would make participation hazardous (e.g., acute, psychosis, current suicidality, current manic episode)
* Has an active, unmanaged medical condition that would make participation hazardous or preclude use of buprenorphine or ancillary medications for withdrawal (e.g., unmanaged hypertension, unmanaged diabetes, clinically significant abnormality on ECG, acute hepatitis)
* Buprenorphine or methadone treatment in the past 30 days
* Known allergy, hypersensitivity or intolerance to buprenorphine
* Pregnancy, lactation, or unwillingness to use adequate contraceptive methods
* Current physiological dependence on sedative-hypnotics or alcohol that would require medically supervised detoxification
* Liver function tests > 2x the upper limit of normal
* Use of medications or herbal products with known CYP3A4 inhibition or induction properties in the past 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Days Abstinent from Opioids | 4 week follow up period
  Abstinence from Opioids (% days abstinent; continuous; longitudinal) during each week of the 4 week follow up period measured via the timeline follow back.
Sustained Relapse | 4 week follow up period
  Sustained relapse during the 4 week follow up period (binary), defined as 5 consecutive days of illicit opioid use reported on the timeline follow back at any point during the 4 week follow up period.

SECONDARY OUTCOMES:
Time to Peak Clinical Opiate Withdrawal Scale (COWS) score | During the inpatient induction period (approximately 1 overnight stay)
  The time to peak Clinical Opiate Withdrawal Scale (COWS) score during the induction period (time-to-event/survival). The COWS ranges from 0-48 with higher scores indicating more severe opioid withdrawal symptoms.
Peak Clinical Opiate Withdrawal Scale (COWS) score | During the inpatient induction period (approximately 1 overnight stay)
  The peak Clinical Opiate Withdrawal Scale (COWS) score during the induction period (continuous). The COWS ranges from 0-48 with higher scores indicating more severe opioid withdrawal symptoms.
Dropout during induction | During the inpatient induction period (approximately 1 overnight stay)
  Dropout during the induction period (binary)

OTHER OUTCOMES:
Exploratory Outcome 1: Craving | Induction Period (Overnight Inpatient Stay) and 4-week follow up period
  Craving as reported on the Opioid Craving Visual Analog Scale OC-VAS (longitudinal; continuous) during induction and follow up. The OC-VAS ranges from 0-100mm with higher ratings indicating more intense/severe craving.
Exploratory Outcome 2: Clinical Opiate Withdrawal Scale (COWS) Score | Induction Period (Overnight Inpatient Stay) and 4-week follow up period
  Opioid Withdrawal Symptoms as reported on the Clinical Opiate Withdrawal Scale (COWS; longitudinal; continuous) during induction and follow up. The COWS ranges from 0-48 with higher scores indicating more severe opioid withdrawal symptoms.
Exploratory Outcome 3: Time to first use of illicit opioids | 4-week follow up period
  Time to first use of illicit opioids during the 4-week follow up period (time-to-event/survival)

CONTACTS AND LOCATIONS:
Locations (1):
- Substance Treatment and Research Service, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
According to NIDA's policy for data management and sharing, de-identified data will be deposited into the NAHDAP repository.
Time Frame: De-identified data will be made available no later than when the primary outcome paper is published or when the award ends. The data will be stored in the repository for at least 10 years after the funding period ends.
Access Criteria: Once released to the repository, the investigator will not control data access.